CLINICAL TRIAL: NCT02736162
Title: A Retrospective Multicenter Study to Investigate Dosage, Efficacy, and Safety of Perampanel Given as Monotherapy in Routine Clinical Care in Patients With Epilepsy
Brief Title: Study to Investigate Dosage, Efficacy, and Safety of Perampanel Given as Monotherapy in Patients With Epilepsy
Status: Completed | Type: Observational
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: E2007-G000-504
Record Dates: First submitted 2016-03-30; First posted 2016-04-13 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Epilepsy; Partial-Onset Seizures; Primary Generalized Tonic-Clonic Seizures
Keywords: Perampanel; E2007; Phase 4; Fycompa
MeSH Terms: conditions — Epilepsy | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Perampanel: Participants with a diagnosis of epilepsy who received perampanel as primary or secondary (conversion) monotherapy at any time between 1 Jan 2013 and 15 Oct 2015.
  Interventions: Other: No treatment (intervention) was administered

INTERVENTIONS:
Other: No treatment (intervention) was administered

SUMMARY:
The primary objective of this study is to assess the retention rate of perampanel when given as secondary monotherapy in routine clinical care.

DETAILED DESCRIPTION:
This study is a retrospective study of participants who received perampanel as primary or secondary monotherapy at approximately 40 centers in Europe, Asia, and Australia. Primary monotherapy is defined as the administration of perampanel in the absence of any concomitant antiepileptic drugs (AEDs). Secondary (conversion) monotherapy is defined as the conversion of perampanel from adjunctive therapy to monotherapy by withdrawing concomitant AEDs.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of epilepsy
* Received perampanel as primary or secondary monotherapy at any time between 1 Jan 2013 and 15 Oct 2015
* Provided written informed consent by the participant or the participant's legally authorized representative signed for the use of medical records per local requirements

Exclusion Criteria:

* Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who received perampanel as primary or secondary monotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2016-04; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Retention rate | Month 3
  The percentage of participants remaining on perampanel monotherapy treatment after conversion from perampanel adjunctive therapy
Retention rate | Month 6
  The percentage of participants remaining on perampanel monotherapy treatment after conversion from perampanel adjunctive therapy
Retention rate | Month 12
  The percentage of participants remaining on perampanel monotherapy treatment after conversion from perampanel adjunctive therapy
Retention rate | Month 18
  The percentage of participants remaining on perampanel monotherapy treatment after conversion from perampanel adjunctive therapy
Retention rate | Month 24
  The percentage of participants remaining on perampanel monotherapy treatment after conversion from perampanel adjunctive therapy
Participants remaining on perampanel monotherapy (after conversion from perampanel as adjunctive therapy) | Up to approximately 34 months

SECONDARY OUTCOMES:
Percentage of participants receiving perampanel monotherapy out of the total number of participants prescribed perampanel | Up to approximately 34 months
Percentage of participants with greater than or equal to 50% reduction in seizure frequency | Up to approximately 34 months
Percentage of participants who were seizure-free for at least 3 months | Up to approximately 34 months
  Seizure-free is defined as a terminal remission of seizures
Percentage of participants with greater than or equal to 75% reduction in seizure frequency | Up to approximately 34 months
Percentage of participants with categorized percent reductions in seizure frequency | Up to approximately 34 months
Percentage of participants with no change or worsening of seizures | Up to approximately 34 months
Median percent change in seizure frequency | Up to approximately 34 months
Percentage of participants with treatment emergent adverse events (TEAEs) and treatment emergent serious adverse events (SAEs) | Up to approximately 34 months
Mean change in body weight | Up to approximately 34 months
Maximum dose of perampanel during adjunctive therapy and monotherapy | Up to approximately 34 months
Average dose of perampanel during adjunctive therapy and monotherapy | Up to approximately 34 months

CONTACTS AND LOCATIONS:
Overall Officials: Karen Cartwright, PhD, Study Director — Eisai Limited